CLINICAL TRIAL: NCT04016246
Title: Respiratory Effect of the LISA (Less Invasive Surfactant Administration) Method with Sedation by Propofol Versus Absence of Sedation: Double-blind Comparative Randomized Clinical Trial.
Brief Title: Respiratory Effect of the LISA Method with Sedation by Propofol Versus Absence of Sedation.
Acronym: PROLISA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC18.123
Record Dates: First submitted 2019-06-07; First posted 2019-07-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: LISA; propofol; medialipide; ketamin; sedation; premature infant; surfactant
MeSH Terms: conditions — Premature Birth | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Experimental): Propofol (Propofol LIPURO 1% 100mL), Pharmacologic form: 10mg/ml. Considering the birthweight of most preterm babies, Propofol will be diluted to a final concentration of 1mg/ml by the nurse.
  Treatment initiation: the 1st dose will be injected following usual management of LISA procedure included the installation of the newborn and the atropine and caffeine injections and sugar solution administration Dose per administration: 0.5mg/kg per dose of Propofol. Number of administrations: Several administrations of 0.5 mg/kg are possible, according the level of sedation achieved, as evaluated by the FANS score. If the FANS score is ≥6, a new dose will be injected up to a total of two (before 28 wGA) or 3 (between 28 - 31 wGA) administrations of the drug. (See paragraph 5.3)
  Interventions: Drug: Propofol-Lipuro
- medialipide (Placebo Comparator): Name of treatment for placebo: Medialipide® (B. BRAUN) Pharmacological form: 20g/100ml Medialipide 20% will be used as the placebo. This is an emulsion of medium and long triglycerides based on soya oil and having same appearance organoleptic characteristics as Propofol.
  Dose per administration: Same volume as for the Propofol administration
  Number of administrations: according the same protocol that for the Propofol administration.
  Modalities of preparation : The same dilution procedure as Propofol lipuro 1% SPC (Summary of Product Characteristics):1 part of Medialipide 20% with 9 parts of 5% w/v glucose solution or 0.9% w/v sodium chloride solution as shown in parenteral nutrition which is in accordance with medialipide 20% SPC
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Propofol-Lipuro — sedation of babies < 32wGA with propofol / placebo before a LISA Procedure
  Arms: Propofol
Drug: Placebos — injected to babies < 32wGA with propofol / placebo before a LISA Procedure
  Other Names: medialipide
  Arms: medialipide

SUMMARY:
The investigators propose to evaluate premedication with Propofol compared to a control strategy including a placebo with a possible rescue treatment with ketamine to ensure pain control before LISA Procedure . Investigators hypothesize that sedation with Propofol is safe and non-inferior to placebo for the risk of Mechanical Ventilation in the 72 hours following the procedure.

DETAILED DESCRIPTION:
Non-inferiority trial comparing Propofol versus placebo during the intra tracheal Less Invasive Surfactant Administration (LISA) in preterm babies < 32 weeks of gestation for the need for mechanical ventilation after the procedure. An open-label ketamine treatment as rescue is possible in each group.

In each participating unit, information will be given to parents of preterm babies <32 wGA upon their admission to the delivery room or to the NICU (neonatal intensive care unit), and informed consent will be sought as soon as possible. Eligible babies presenting a RDS (respiratory distress syndrome) will be included and randomized to the control (placebo) group or Propofol group. While benefiting from Nasal Intermittent Positive Pressure Ventilation (NIPPV) the newborn will be prepared as usual for tracheal intubation. Trialists will be blinded to treatment allocation.

The drug administration in the two groups will be titrated according to weight (0.5mg/kg per dose of Propofol or a similar volume of placebo). After each dose, a pain score (FANS) will be quickly evaluated within 2 minutes of the injection, to assess the need for a supplementary dose (up to a predefined limit) or rescue treatment by Ketamine.

After the steps of sedation, the LISA procedure will be performed, with detailed data collection of per procedure events up to 72 hours of life. Babies will be subsequently managed as usual in each NICU and data will be collected about respiratory, neurological and hemodynamic outcomes during the hospital stay, and especially at discharge, 28 days, and 36 weeks. At two years of corrected age, a final examination will be performed to evaluate neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants < 32 wGA (weeks of gestational age)
* Presenting a RDS (respiratory distress syndrome)

  * in the first 48 hours of life
  * treated by CPAP (continuous positive airway pressure) or BiPAP (Bilevel Positive Airway Pressure)
  * requiring surfactant :

    * FIO2 : (fraction of inspired oxygen)

      * if 28 - 31 SA : FiO2 ≥30% for a duration ≥ 10mn
      * if <28 SA FIO2 ≥25% for a duration ≥10mn
    * SpO2 (arterial oxygen saturation) : to obtain a SpO2 between ≥88 and ≤ 95%
* Available IntraVenous line (peripheral, umbilical or central catheter)
* Recipient of the French Social Security
* Informed consent form signed

Exclusion Criteria:

* Congenital and/or major malformations
* FIO2 >60%
* Silverman score >6
* Contraindication to the use of Propofol :
* Low Blood Pressure with 2 successive measurements (Mean < Gestational Age expressed in Weeks of Gestation) persisting after one volume expansion,
* Use of inotropic medication to maintain a normal blood pressure.
* Use of sedative or analgesic drugs (except paracetamol and ibuprofen) in the previous 24h
* Coma, convulsions, areactivity at neurological examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
need for mechanical ventilation after the procedure | 72hours
  Rate of mechanical ventilation from the start of the LISA procedure up to 72 hours of life.

SECONDARY OUTCOMES:
Rate of MV (mechanical ventilation ) in each class of GA (<28, 28-31wGA) | 72hours
  Rate of MV (mechanical ventilation
  ) from the start of the LISA procedure up to 72 hours of life in each class of GA (<28, 28-31wGA)
FANS during LISA and 1h after LISA | 1hour
  Faceless acute neonatal pain scale (FANS) assessed during LISA and 1 hour after the procedure by an independent operator.
number of ketamine administrations for rescue | before LISA Procedure
  Number of ketamine administrations for rescue in order to obtain a FANS score <6 and to be able to proceed to LISA.
Number of laryngoscopies | during LISA Procedure (T0)
  Number of laryngoscopies needed to perform LISA
Tolerance and efficacy (Per procedure events): Apnea | during LISA Procedure (T0)
  Apnea requiring bag mask ventilation
Tolerance and efficacy (Per procedure events): emergency intubation | from drug injection to 1hour after
  Emergency intubation after the drug injection before the LISA procedure can be performed or within 1h following the drug injection
Tolerance and efficacy (Per procedure events): Viby Mogensen score | during LISA Procedure
  Clinician's satisfaction during laryngoscopy with the Viby Mogensen score :
  Item Score 1 Score 2 Score 3 Score 4 Laryngoscopy Easy Fair Difficult Impossible Vocal cords Open Moving Closing Closed Coughing None Slight Moderate Severe Jaw relaxation Complete Slight Stiff Rigid Limb movements None Slight Moderate Severe
  the total score is calculated adding each item scores. min score = 5. max score = 20. An easy intubation would obtain a low score and a difficult intubation would have a high score.
BPD (bronchopulmonary dysplasia) at 36 weeks of Gestational Age | equivalent to 36 weeks of Gestational Age
  Broncho Pulmonary Dysplasia at 36 weeks of Gestational Age
In-hospital morbidity and mortality: pneumothorax | 72hours post LISA Procedure
  Pneumothorax within 72hours
In-hospital morbidity and mortality: Necrotizing Enterocolitis | the day of discharge from hospital (the day depends to each participant : between 36-45 weeks of Gestational Age)
  necrotizing enterocolitis during hospitalization
In-hospital morbidity and mortality : sepsis | the day of discharge from hospital (the day depends to each participant : between 36-45 weeks of Gestational Age)
  proven sepsis during hospitalization
In-hospital morbidity and mortality: retinopathy | the day of discharge from hospital (the day depends to each participant : between 36-45weeks of gestational ageGA)
  retinopathy of prematurity during hospitalization
In-hospital morbidity and mortality | the day of discharge from hospital (the day depends to each participant : between 36-45weeks of Gestational Age)
  periventricular leukomalacia or grade 3 or 4 intraventricular hemorrhage during hospitalization
In-hospital morbidity and mortality: patent ductus arteriosus | the day of discharge from hospital (the day depends to each participant : between 36-45 weeks of Gestational Age)
  treatment of a patent ductus arteriosus during hospitalization
In-hospital morbidity and mortality: death 36weeks of Gestational Age | equivalent to 36 weeks of Gestational Age
  Death at 36 weeks of Gestational Age
In-hospital morbidity and mortality: death during hospitalization | the day of discharge from hospital (the day depends to each participant : between 36-45weeks of Gestational Age)
  in-hospital mortality
At two years of corrected age: ASQ (Ages and Stages Questionnaire) | 2 years (corrected age)
  ASQ (Ages and Stages Questionnaire) questionnaire is a general developmental screening tool (5 areas are evaluated: Communication, gross motor, fine motor, problem solving, and personal-social). Total score is the sum of each of the 5 area scores (wich are between 0-60. Total score is between 0 and 300. The higher the score is, the best developed the children is.
At two years of corrected age: motor function | 2 years (corrected age)
  Gross Motor Function Classification Scale (GMFCS) looks at movements such as sitting, walking and use of mobility devices. It is helpful because it provides families and clinicians with a clear description of a child's current motor function, and an idea of what equipment or mobility aids a child may need in the future, e.g. crutches, walking frames or wheelchairs.
  Participant will be assignated to one of the 5 levels by the clinicians : a patient who is in level 5 has more motor impairments than a patient in level 1.
At two years of corrected age: vision | 2 years (corrected age)
  Visual functions : a clinical examination will conclude if the participant has a visual deficit or not. And in the deficit case, what kind of vision pathology.
At two years of corrected age: audition | 2 years (corrected age)
  Hearing functions : a clinical examination will conclude if the participant has a hearing deficit or not. And in the deficit case, what kind of audition pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DEBILLON, MD PHD, Principal Investigator — CHU de Grenoble Alpes
Locations (13):
- France (13):
  - centre hospitalier deTroyes, Troyes, aube
  - CHU Grenoble Alpes, Grenoble, Isère
  - Chu Amiens, Amiens
  - Chu Angers, Angers
  - Chu Brest, Brest
  - Chu Chambery, Chambéry
  - Chi Creteil, Créteil
  - Chu Limoges, Limoges
  - Ap-H Marseille, Marseille
  - Chu Nantes, Nantes
  - Chu Nimes, Nîmes
  - Chi Poissy St Germain, Poissy
  - Ch Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dekker J, Lopriore E, Rijken M, Rijntjes-Jacobs E, Smits-Wintjens V, Te Pas A. Sedation during Minimal Invasive Surfactant Therapy in Preterm Infants. Neonatology. 2016;109(4):308-13. doi: 10.1159/000443823. Epub 2016 Feb 24. PMID 26907795
- [Background] Dargaville PA, Kamlin CO, De Paoli AG, Carlin JB, Orsini F, Soll RF, Davis PG. The OPTIMIST-A trial: evaluation of minimally-invasive surfactant therapy in preterm infants 25-28 weeks gestation. BMC Pediatr. 2014 Aug 27;14:213. doi: 10.1186/1471-2431-14-213. PMID 25164872
- [Background] Gopel W, Kribs A, Ziegler A, Laux R, Hoehn T, Wieg C, Siegel J, Avenarius S, von der Wense A, Vochem M, Groneck P, Weller U, Moller J, Hartel C, Haller S, Roth B, Herting E; German Neonatal Network. Avoidance of mechanical ventilation by surfactant treatment of spontaneously breathing preterm infants (AMV): an open-label, randomised, controlled trial. Lancet. 2011 Nov 5;378(9803):1627-34. doi: 10.1016/S0140-6736(11)60986-0. Epub 2011 Sep 29. PMID 21963186
- [Background] Dekker J, Lopriore E, van Zanten HA, Tan RNGB, Hooper SB, Te Pas AB. Sedation during minimal invasive surfactant therapy: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F378-F383. doi: 10.1136/archdischild-2018-315015. Epub 2018 Aug 1. PMID 30068669
- [Background] Berde CB, Walco GA, Krane EJ, Anand KJ, Aranda JV, Craig KD, Dampier CD, Finkel JC, Grabois M, Johnston C, Lantos J, Lebel A, Maxwell LG, McGrath P, Oberlander TF, Schanberg LE, Stevens B, Taddio A, von Baeyer CL, Yaster M, Zempsky WT. Pediatric analgesic clinical trial designs, measures, and extrapolation: report of an FDA scientific workshop. Pediatrics. 2012 Feb;129(2):354-64. doi: 10.1542/peds.2010-3591. Epub 2012 Jan 16. PMID 22250028
- [Background] Bourgoin L, Caeymaex L, Decobert F, Jung C, Danan C, Durrmeyer X. Administering atropine and ketamine before less invasive surfactant administration resulted in low pain scores in a prospective study of premature neonates. Acta Paediatr. 2018 Jul;107(7):1184-1190. doi: 10.1111/apa.14317. Epub 2018 Apr 16. PMID 29532502
- [Background] Ghanta S, Abdel-Latif ME, Lui K, Ravindranathan H, Awad J, Oei J. Propofol compared with the morphine, atropine, and suxamethonium regimen as induction agents for neonatal endotracheal intubation: a randomized, controlled trial. Pediatrics. 2007 Jun;119(6):e1248-55. doi: 10.1542/peds.2006-2708. Epub 2007 May 7. PMID 17485450
- [Background] Owen LS, Manley BJ. Nasal intermittent positive pressure ventilation in preterm infants: Equipment, evidence, and synchronization. Semin Fetal Neonatal Med. 2016 Jun;21(3):146-53. doi: 10.1016/j.siny.2016.01.003. Epub 2016 Feb 26. PMID 26922562
- [Background] Durrmeyer X, Daoud P, Decobert F, Boileau P, Renolleau S, Zana-Taieb E, Saizou C, Lapillonne A, Granier M, Durand P, Lenclen R, Coursol A, Nicloux M, de Saint Blanquat L, Shankland R, Boelle PY, Carbajal R. Premedication for neonatal endotracheal intubation: results from the epidemiology of procedural pain in neonates study. Pediatr Crit Care Med. 2013 May;14(4):e169-75. doi: 10.1097/PCC.0b013e3182720616. PMID 23439457
- [Background] Kanmaz HG, Erdeve O, Canpolat FE, Mutlu B, Dilmen U. Surfactant administration via thin catheter during spontaneous breathing: randomized controlled trial. Pediatrics. 2013 Feb;131(2):e502-9. doi: 10.1542/peds.2012-0603. Epub 2013 Jan 28. PMID 23359581
- [Background] Descamps CS, Chevallier M, Ego A, Pin I, Epiard C, Debillon T. Propofol for sedation during less invasive surfactant administration in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F465. doi: 10.1136/archdischild-2017-312791. Epub 2017 May 8. No abstract available. PMID 28483817
- [Background] Klotz D, Porcaro U, Fleck T, Fuchs H. European perspective on less invasive surfactant administration-a survey. Eur J Pediatr. 2017 Feb;176(2):147-154. doi: 10.1007/s00431-016-2812-9. Epub 2016 Dec 9. PMID 27942865
- [Derived] Chevallier M, Durrmeyer X, Ego A, Debillon T; PROLISA Study Group. Propofol versus placebo (with rescue with ketamine) before less invasive surfactant administration: study protocol for a multicenter, double-blind, placebo controlled trial (PROLISA). BMC Pediatr. 2020 May 8;20(1):199. doi: 10.1186/s12887-020-02112-x. PMID 32384914